CLINICAL TRIAL: NCT00090623
Title: A Phase IIIb, Multicenter, Randomized, Double Masked, Sham Injection-Controlled Study of the Efficacy and Safety of Ranibizumab in Subjects With Subfoveal Choroidal Neovascularization (CNV) With or Without Classic CNV Secondary to Age Related Macular Degeneration
Brief Title: A Study of rhuFab V2 (Ranibizumab) in Subjects With Subfoveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FVF3192g
Record Dates: First submitted 2004-08-30; First posted 2004-09-01 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Macular Degeneration
Keywords: Subfoveal neovascular; Age-related macular degeneration; AMD; Wet AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

INTERVENTIONS:
Drug: rhuFab V2 (ranibizumab)

SUMMARY:
This is a phase III, multicenter, randomized, double masked, sham injection-controlled study of the efficacy and safety of intravitreally administered ranibizumab in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >=50 years
* Active primary or recurrent subfoveal CNV lesions secondary to AMD in the study eye
* Total area of CNV (including both classic and occult components) encompassed within the lesion >= 50% of the total lesion area
* Total lesion area <=12 disc areas in size
* Best corrected visual acuity (BCVA), using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts, of 20/40 to 20/320 (Snellen equivalent) in the study eye

Exclusion Criteria:

* Prior treatment with verteporfin, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* Treatment with verteporfin in the nonstudy eye <7 days preceding Day 0
* Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)
* Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Day 0
* History of vitrectomy surgery in the study eye
* History of submacular surgery or other surgical intervention for AMD in the study eye
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)
* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either >= 50% of the total lesion area or >=1 disc area in size
* Fibrosis or atrophy involving the center of the fovea in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either: (1) Require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition, or (2) If allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 24-month study period
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >=30 mmHg despite treatment with antiglaucoma medication)
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Premenopausal women not using adequate contraception
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded by the central reading center
* Inability to comply with study or follow up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-08; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Trial Information Support Line, Denver, Colorado, United States

REFERENCES:
- [Result] Regillo CD, Brown DM, Abraham P, Yue H, Ianchulev T, Schneider S, Shams N. Randomized, double-masked, sham-controlled trial of ranibizumab for neovascular age-related macular degeneration: PIER Study year 1. Am J Ophthalmol. 2008 Feb;145(2):239-248. doi: 10.1016/j.ajo.2007.10.004. PMID 18222192
- [Derived] Barbazetto I, Saroj N, Shapiro H, Wong P, Freund KB. Dosing regimen and the frequency of macular hemorrhages in neovascular age-related macular degeneration treated with ranibizumab. Retina. 2010 Oct;30(9):1376-85. doi: 10.1097/IAE.0b013e3181dcfb0b. PMID 20683380
- [Derived] Abraham P, Yue H, Wilson L. Randomized, double-masked, sham-controlled trial of ranibizumab for neovascular age-related macular degeneration: PIER study year 2. Am J Ophthalmol. 2010 Sep;150(3):315-324.e1. doi: 10.1016/j.ajo.2010.04.011. Epub 2010 Jul 3. PMID 20598667